CLINICAL TRIAL: NCT07246239
Title: Evaluating the Effectiveness of an Online Cognitive Behavioral Therapy Program for University Students With Depression and/or Anxiety: A Randomized Controlled Trial
Brief Title: Evaluating the Effectiveness of an Online Cognitive Behavioral Therapy Program for University Students With Depression and/or Anxiety
Acronym: VIVIM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Rovira i Virgili (Other)
Collaborators: University Ramon Llull (Other); Universitat de Girona (Other)
Responsible Party: Principal Investigator, Anna Huguet, PhD, University Rovira i Virgili
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEIPSA-2024-PR-0023 Full RCT; 2023 Benes 00023 (Other Grant/Funding Number: Agència de la Gestió d'Ajuts Universitaris i de Recerca (AGAUR))
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Anxiety and Depression
Keywords: cognitive-behavioral treatment; internet-based program; depression; anxiety; students; university
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Counseling

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet-based CBT program (Experimental): This 10-week program consists of 10 modules. Throughout the program, participants progress at their own pace. They have the opportunity to attend two individual support sessions (at the beginning and midway through the program) as well as in weekly group support designed to address questions and reinforce learning. These sessions are conducted via videoconference. Participants also receive weekly automated email remainders and can contact the team via email at any time.
  This program is an adaptation of Overcoming Low mood and Depresion: A Five Areas Approach.
  Interventions: Behavioral: VIVIM (Viure la Vida al Màxim/Vivir la Vida al Máximo)
- Treatment as usual (Active Comparator): Treatment as usual involves referral to the counseling service offered by the university to its students.
  Interventions: Other: Counseling

INTERVENTIONS:
Behavioral: VIVIM (Viure la Vida al Màxim/Vivir la Vida al Máximo) — This is the Internet-based CBT program
  Arms: Internet-based CBT program
Other: Counseling — This is the type of support that is offered from the university counseling services
  Arms: Treatment as usual

SUMMARY:
The goal of this clinical trial is to learn if an Internet-based self-help program called VIVIM can help university students with depression and/or anxiety. The main question we want to answer is:

* Does the VIVIM program help participants to feel less depressed and/or anxious? We will compare the VIVIM program with the usual psychological support that university counselling services offer to students.

Participants will:

* Be randomly assigned to either use the VIVIM program or receive usual help from university's counselling service.
* Fill out online questionnaires three times: at the beginning, 10 weeks and 6 months after being assigned either the VIVIM program or usual care.

ELIGIBILITY:
Inclusion Criteria:

* To be enrolled as an undergraduate or postgraduate at of the participating Spanish universities.
* To report at least moderate symptoms of depression (PHQ>o= 10) and/or anxiety (GAD-7>o= 10).

Exclusion Criteria:

* To self-report having been diagnosed with bipolar and/or psychotic disorder.
* To report to be currently receiving psychotherapy/counselling and/or pharmacological treatment for emotional problems.
* To be unable to read, speak or understand Spanish.
* To be at risk of suicide.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Anxiety | From enrollment to 6 months after being randomized
  The Generalized Anxiety Disorder [GAD-7] will be used
Depression | From enrollment to 6 months after being randomized
  The Patient Health Questionnaire-9 item [PHQ-9] will be used

SECONDARY OUTCOMES:
Functional impairment | From enrollment to 6 months after being randomized
  Work and Social Adjustment Scale [WSAS] will be used
Mental well-being | From enrollment to 6 months after being randomized
  The Five Well-Being Index will be used
Resilience | From enrollment to 6 months after being randomized
  The Connor-Davidson Resilience Scale [CD-RISC-10] will be used

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - Blanquerna - Universitat Ramon Llull, Barcelona, Barcelona
  - Universitat de Girona, Girona, Girona
  - Universitat Rovira i Virgili, Tarragona, Tarragona

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in a publication will be shared in the data repository of the Univesitat Rovira i Virgili.
Time Frame: Starting 6 months after publication with no end date.